CLINICAL TRIAL: NCT06666244
Title: Evaluation of the Effect of Carbohydrate Quality on Quality of Life and Menopausal Symptoms in Postmenopausal Women
Brief Title: Carbohydrate Quality, Quality of Life, and Menopausal Symptoms in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assist Prof, Ankara Yildirim Beyazıt University
Other Study IDs: AYBUELİBOL004
Record Dates: First submitted 2024-10-23; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-09

CONDITIONS: Woman
Keywords: Carbohydrate Quality; Quality of life; Menopausal Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Postmenopausal Women: This study aimed to evaluate the effect of carbohydrate quality on quality of life and menopausal symptoms in postmenopausal women. Data were collected from 604 postmenopausal women using a demographic questionnaire, the Menopause-Specific Quality of Life Questionnaire (MENQOL), and the Menopause Rating Scale (MRS). Carbohydrate quality was assessed using food frequency consumption data, and results were analyzed with SPSS 24 software.

SUMMARY:
This study aimed to evaluate the effect of carbohydrate quality on quality of life and menopausal symptoms in postmenopausal women. Data were collected from 604 postmenopausal women using a demographic questionnaire, the Menopause-Specific Quality of Life Questionnaire (MENQOL), and the Menopause Rating Scale (MRS). Carbohydrate quality was assessed using food frequency consumption data, and the results were analyzed with SPSS 24 software.

DETAILED DESCRIPTION:
Objective: This study aimed to evaluate the effect of carbohydrate quality on quality of life and menopausal symptoms in postmenopausal women.

Method: A total of 604 postmenopausal women participated in the study. Participants completed a demographic questionnaire, the Menopause-Specific Quality of Life Questionnaire (MENQOL), and the Menopause Rating Scale (MRS). Carbohydrate quality was assessed using food frequency consumption data and analyzed based on dietary fiber, glycemic index, solid carbohydrate-to-total carbohydrate ratio, and whole grains-to-total grains ratio. Results were divided into five quartiles, with Q5 representing the highest and Q1 the lowest carbohydrate quality. Data analysis was conducted using SPSS 24 software.

ELIGIBILITY:
Inclusion Criteria:

* Women who have not menstruated for 12 consecutive months and have no intermenstrual bleeding
* Aged between 30 and 90 years
* Must be willing to volunteer

Exclusion Criteria:

* Women diagnosed with any psychological disorder
* Cancer patients

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample in Ankara, Turkey
Sampling Method: Probability Sample
Enrollment: 604 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluating carbohydrate quality | Basaline
  132 food groups obtained from the food consumption frequency questionnaire were analyzed. Daily intake (g/day) was calculated using the BeBiS program with a global database, based on the amount and frequency of food consumed by participants. Glycaemic Index (GI) values were also determined using the BeBiS program, taking into account both the amount and frequency of food consumed. To determine the Carbohydrate Quality Index score, each of the four components (fiber intake, whole grain ratio, Glycaemic Index, and total carbohydrate ratio) was rated from 1 to 5 points. The score for each component was then summed. Q5 indicates the highest and Q1 the lowest carbohydrate quality.

SECONDARY OUTCOMES:
Menopause-Specific Quality of Life Questionnaire (MENQOL) | Basaline
  This scale is used to assess quality of life during menopause. It consists of 29 questions across four subdimensions, with scores ranging from 1 to 8. Higher scores on this scale indicate greater severity of complaints.
Menopause Rating Scale (MRS) | Basaline
  This scale was used to measure the severity and frequency of menopausal symptoms. It includes three subdimensions: psychological, somatic, and urogenital complaints. Each question has five response options (scored from 0 to 4), with a total possible score of 44 and a minimum score of 0. Higher scores indicate a greater negative impact on quality of life and an increase in symptoms.
Sociodemographic characteristics | Basaline
  Sociodemographic characteristics will be assessed using a structured questionnaire developed by the researchers. The questionnaire will include items on age, gender, education level, and income status. Results will be presented as frequencies and percentages for each characteristic.
Body Mass Index (BMI) | Basaline
  Kilograms per square meter (kg/m2)
Body weight | Basaline
  Body weight in kg
Height | Basaline
  Height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No